CLINICAL TRIAL: NCT03413007
Title: Correlation Between Immune compleX Predictive Index and Prostate Cancer Aggressiveness at Radical Prostetecomy Specimens: a Multicenter Prospective Trial
Brief Title: Correlation Between iXip and Final Pathology Specimen From Radical Prostatectomy: a Multicenter Prospective Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alessandro Antonelli, Urology consultant, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: PSA-IgM
Record Dates: First submitted 2018-01-16; First posted 2018-01-29 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — a blood serum sample will be stored for each patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immune compleX Predictive Index — iXip is an algorithm thant integrates PSA, PSA-IgM, prostate volume and age of the patient in order to provide the probability of prostate cancer

SUMMARY:
The Immune compleX Predictive Index (iXip) is a predictive tool for prostate cancer (PCa) diagnosis that integrates PSA, PSA-IgM, prostate volume and age of the patient. An algorithm processes these parameters providing the probability of prostate cancer. Several prospective studies confirmed its ability to predict prostate cancer presence at biopsy and therefore to reduce the rate of useless prostate biopsies. Moreover, preliminary results from a prospective study showed that iXip could predict cancer aggressiveness, too.

DETAILED DESCRIPTION:
Since the 90s, serum PSA has become the cornerstone of diagnosis of PCa, However, due to its proven poor specificity, the actual role of PSA testing has been largely debated, especially if used during opportunistic screening programs. leading to a significant risk of over-diagnosis and over treatment.

In order to overcome drawbacks of PSA-based diagnostic pathway several PSA-derivates has been proposed. However, they were marginally used in clinical practice because not supplied by public health care systems.

The Immune compleX Predictive Index (iXip) is a predictive tool for prostate cancer (PCa) diagnosis that integrates PSA, PSA-IgM, prostate volume and age of the patient. An algorithm processes these parameters providing the probability of prostate cancer. Several prospective studies confirmed its ability to predict prostate cancer presence at biopsy and therefore to reduce the rate of useless prostate biopsies. Moreover, preliminary results from a prospective study showed that iXip could predict cancer aggressiveness, too.

All pathological specimens are analyzed by an expert uropathologist, following ISUP reccomandations.

Before radical prostectomy a blood sample from each patients is collected. Serum PSA-IgM concentration is measured using Prostate-IC kit in duplicate. The analysis with Prostate-IC kit was performed on automated ELISA analyzer.Then the iXip index is calculated by using the online calculator (http://ixip.xeptagen.com/).

ELIGIBILITY:
Inclusion Criteria are:

* histologically proven prostate cancer,
* patients scheduled for radical prostatectomy
* paziente able to provide consent
* age > 18 years or < 80 years

Exclusion criteria are:

* neiadjuvant hormone therapy
* salvage radical prostatectomy
* concomitant solid or hematological tumors,
* autoimmune disorders
* or immunosuppressive therapies,
* acute bacterial or viral infections.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male patients with prostate cancer scheduled for radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
correlation between iXip and significant prostate carcer | 6 months after surgery
  correlation between iXip and significant prostate carcer at final pathology specimens, defined as tumor volume > 0.5 cm3 and Gleason scor equal or superior to 7. iXip values are expressed as a percentage and vary from 0% to 100%. Higher iXip values (>30%) should be associated with aggressive pathological features.

SECONDARY OUTCOMES:
correlation between iXip and tumor volume > 0.5 cm3 | 6 months after surgery
  clinical and pathological correlation between iXip values and tumour volume at final pathology specimens. iXip values are expressed as a percentage and vary from 0% to 100%. Higher iXip values (>30%) should be associated with aggressive pathological features ( >0.5cm3 tumor volume )
correlation between iXip and tumor volume > 2.5 cm3 | 6 months after surgery
  clinical and pathological correlation between iXip values and tumour volume at final pathology specimens. iXip values are expressed as a percentage and vary from 0% to 100%. Higher iXip values (>30%) should be associated with aggressive pathological features ( >2.5cm3 tumor volume ).
correlation between iXip and Gleason Score >6 | 6 months after surgery
  clinical and pathological correlation between iXip values and tumour volume at final pathology specimens. iXip values are expressed as a percentage and vary from 0% to 100%. Higher iXip values (>30%) should be associated with aggressive pathological features ( Gleason Score> 6)
correlation between iXip and pathological stage > pT2 | 6 months after surgery
  clinical and pathological correlation between iXip values and tumour volume at final pathology specimens. iXip values are expressed as a percentage and vary from 0% to 100%. Higher iXip values (>30%) should be associated with aggressive pathological features ( pathological staging >pT2)
correlation between iXip and positive lymph node at final pathology specimens | 6 months after surgery
  clinical and pathological correlation between iXip values and tumour volume at final pathology specimens. iXip values are expressed as a percentage and vary from 0% to 100%. Higher iXip values (>30%) should be associated with aggressive pathological features ( positive lymph nodes >0)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Antonelli, Principal Investigator — Spedali Civili Hospital, Brescia (Italy)
Locations (1):
- ASST Spedali Civili of Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided